CLINICAL TRIAL: NCT03984942
Title: Bypass Post-Anesthesia Care Unit(PACU) in Knee and Hip Arthroplasty - A Quality Cohort Study
Brief Title: Bypass PACU in Knee and Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Niklas Ingemann Nielsen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Niklas Ingemann Nielsen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Other Study IDs: NBF_EKAa_01_2019
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Surgery; Knee Osteoarthritis; Postoperative Complications; Hip Osteoarthritis; Arthroplasty Complications
Keywords: Knee Arthroplasty; Hip Arthroplasty; Postoperative Anaesthesia Care Unit
MeSH Terms: conditions — Osteoarthritis, Knee; Postoperative Complications; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Quality Study in the use of Post-Anaesthesia Care Unit(PACU) in Hip and Knee Arthroplasty, and the ability to bypass this unit.

The investigators wish to investigate the amount of patients who is required to be secondary admitted to the PACU, after primary discharge from the operating room to the surgical ward, thereby bypassing the PACU.

DETAILED DESCRIPTION:
The investigators wish to investigate the use of our standardized regimen for discharging patients directly to the surgical ward, thereby bypassing the PACU. The anaesthesiology dept. have a local standard operating procedure for doing this, and the patients will be treated according to this.

This means that Patients will be discharged directly to the surgical ward if the following criteria are met:

* American Society of Anaesthesiologist-score (ASA-score) < 3
* Anaesthesia and surgery without any complications, vital signs normal during the whole procedure and not demanding oxygen supplement on the end of the procedure.
* Bloodloss < 500 ml.
* Postoperative evaluation, Early Warning Score, and postoperative score documented in Electronic Patient journal(EPJ).

The patients will upon arrival at the surgery start a registration containing preoperative data(baseline morbidity, sex, height, weight, type of anaesthesia and surgery), perioperative data containing surgery and anaesthesia data, and postoperative discharge-score(local operating procedure).

After discharge to either the surgical ward or the PACU, the patient will be observed closely the first 2 hours while recording every intervention made by the nurse staff.

After the initial 2 hours the recording goes on the next 24 hours recording every event and intervention which lead to a doctor consult, by telephone or physically examining the patient.

Also, the investigators wish to evaluate the use of the discharge Score(Danish Society of Anaesthesia and Intensive care Medicine(DASAIM)-SCORE), which is used as the discharge score after surgery in other hospitals in Denmark, and the investigators therefore record this after surgery, and every 30 minutes after the surgery for the first 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective unilateral primary Hip- og Knee-Arthroplasty and unicompartmental Knee-Arthroplasty.
* Above 18 years.

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient planned for unilateral Primary Total Hip and Knee Arthroplasty and unilateral unicompartmental knee arthroplasty within a year, or until 600 patients is included.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Bypassing PACU | Within the first 24 hours.
  Number of patients in need of secondary relocation to the Post Anaesthesia Care unit after knee and hip arthroplasty.

SECONDARY OUTCOMES:
Postoperative actions and interventions by nurses within 2 hours. | 2 hours after surgery.
  Postoperative interventions carried out within the first 2 hours after surgery. These interventions will be recorded in a preformed chart.
  The recording will take place booth in the PACU and in the surgical ward, to thereby make a comparison of the two.
Postoperative actions and interventions within 24 hours. | 24 hours after surgery.
  Postoperative interventions and deviant events/complications that require a contact to a medical doctor, either by telephone or personal oversight, carried out within the first 24 hours after surgery.
  These interventions will be recorded in a preformed chart. This registration will take place where the patient is hospitalized at the current timeframe.
30 day Follow-up. | 30 days
  30 day follow-up after surgery, concerning readmission within 8 days after surgery, length of stay and mortality.
90 day Follow-up. | 90 days
  90 day follow-up after surgery concerning readmission and mortality.
Complications after surgery. | 90 days
  Complications after surgery, divided in medical and surgical complications with details of type of event and time of occurence as well as treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eske Aasvang, Dr.Med., Study Director — Centre for abdominal surgery, rigshospitalet.
Locations (1):
- Hvidovre Hospital, Capital Region of Denmark., Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Planned sharing data upon request.